CLINICAL TRIAL: NCT04023591
Title: Nerve Transfers to Improve Upper Extremity Function and Quality of Life in Tetraplegic Patients
Brief Title: Nerve Transfer After Spinal Cord Injury- Multi-center
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Stanford University (Other); University of Pennsylvania (Other); University of Michigan (Other); University of Calgary (Other); University of Utah (Other); United States Department of Defense (U.S. Federal Agency); The Methodist Hospital Research Institute (Other); University of Miami (Other); University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: SC180063
Record Dates: First submitted 2019-07-11; First posted 2019-07-17 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Tetraplegia; Spinal Cord Injuries; Quadriplegia Flaccid
Keywords: tetraplegia; spinal cord injury; quadriplegia; nerve transfer
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries | interventions — Surgical Procedures, Operative; Occupational Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Surgery: Surgery/ Occupational Therapy
  Interventions: Procedure: Surgery/Occupational Therapy

INTERVENTIONS:
Procedure: Surgery/Occupational Therapy — Surgery based on function and injury/ Occupational therapy for 48 months post-surgery

SUMMARY:
Current treatment strategies of acute cervical spinal cord injuries remain limited. Treatment options that provide meaningful improvements in patient quality of like and long-term functional independence will provide a significant public health impact. Specific aim: Measure the efficacy of nerve transfer surgery in the treatment of patients with complete spinal cord injuries with no hand function. Optimize the efficiency of nerve transfer surgery by evaluating patient outcomes in relation to patient selection and quality of life and functional independence.

DETAILED DESCRIPTION:
Study Design and Feasibility: A prospective multi-institutional non-randomized single arm design will be utilized. Seventy subjects with cervical ASIA A-B (International Standards for Neurological Classification of Spinal Cord Injury) SCI and hand function impairment that fit the International Classification for Surgery of the Hand 0-4 will be identified. Only patients with stable ASIA scores and no evidence of functional improvement in motor or sensory examination for at least 3 months will be recruited. All patients will undergo Electromyography (EMG) and nerve conduction studies (NCS) to verify intact innervation (normal compound muscle action potentials (CMAPs)) to the paralyzed target muscles below the level of injury. Functional electrical stimulation (FES) will be used to verify loss of lower motor neuron function in key muscle groups in the zone of injury and help differentiate those muscle with intact connections to preserve anterior horn cells. Only those patients with clinically normal, Medical Research Council (MRC) muscle grade 5/5 donor (axonal donor) function will be enrolled.

Outcome Measures Primary Outcome Measures: Pre- and Post-operative upper motor strength. (Manual motor testing & Hand Held Dynamometry) Secondary Outcome Measures: Disabilities of the Arm, Shoulder, and Hand (DASH), Michigan Hand Questionnaire (MHQ), Spinal Cord Injury Quality of Life (SCIQOL), GRASSP test (pre-operative, post-operatively - 6 months, 12 months, and 24 months, 36 months and 48 months), rates of intraoperative and post-operative complications, and rates of reoperation.

Rehabilitation and hand therapy are critical components of motor re-education following nerve transfers. Cortical plasticity and motor remapping occurs following nerve transfers allowing independent functional control of the recipient muscles. All patients will begin rehabilitation and hand therapy beginning 2 weeks after surgery. They undergo one hour of hand therapy and occupational therapy for motor re-education once to twice a week for 48 months following surgery. Rehabilitation will be phased to early and late - added exercises focusing on co-contraction, repetition, and range of motion will be included as home therapy.

ELIGIBILITY:
Inclusion Criteria

1. Age 18-65, inclusive
2. At least 3 months of non-operative rehab therapy
3. Mentally and physically willing and able to comply with evaluations
4. Less than 36 months post-injury
5. Stable ASIA scores with no evidence of functional improvement in motor or sensory examination for at least 3 months
6. ASIA A or B determined by the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI)
7. EMG/NCS verifies intact innervation (normal CMAPs) to the paralyzed target muscles below the level of injury
8. Functional electrical stimulation (FES) will be performed. Subject must have clinically normal MRC grade 5/5 donor (axonal) function
9. Injury Level C4-C8

Exclusion Criteria

1. Active infection at the operative site or systemic infection
2. Any return or ongoing clinical recovery of distal motor function
3. Mentally or physically compromised that will prevent them from complying with evaluations.
4. Immunologically suppressed
5. Currently undergoing long-term steroid therapy
6. Active malignancy
7. Pregnant
8. Significant joint contractures and/or limitations in passive range of motion in the arm or hand, per treating surgeon's discretion
9. Lack of appropriate social support and/or infrastructure to commit to scheduled follow-up visits.
10. Patients who are planning on undergoing a tendon transfer during the study period or who have had a tendon transfer in the past.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a traumatic cervical spine injury with little to no use of his/her arms/hands.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Manual Motor Testing | 48 months
  Change from baseline testing strength of upper extremities at 48 months post-operatively
Handheld Dynamometry | 48 months
  Change from baseline grip strength at 48 months post-operatively

SECONDARY OUTCOMES:
Change in Disabilities of Arm, Shoulder and Hand (DASH) scores | 48 months
  Change from baseline DASH scores at 48 months post-operatively. Scores range from 0-100 with 0 being the most positive score representing no arm, shoulder or hand disability and 100 being the lowest score indicating the most severe arm, shoulder and hand disability.
Change in Spinal Cord Injury Quality of Life (SCIQOL) scores | 48 months
  Change in baseline SCIQOL scores at 48 months post-operatively. Five scores of 0-30 (0=less satisfied and 30=most satisfied) are calculated: 1. Total Quality of Life; 2. Health and Functioning Subscale; 3. Social and Economic Subscale; 4. Psychological/Spiritual Subscale; 5 Family Subscale. Calculation of scores weighs satisfaction scores according to level of importance assigned to each item. An overall score can be obtained by summing the scores for all six scales after reversing the pain scale and dividing by six.
Rates of Intra-operative and post-operative complications | 48 months
  The number of complications within and after the operation
Hand Function, measured by the GRASSP test | 48 months
  Change in baseline GRASSP Test results for hand function at 48 months post-operatively
Changes in the Graded Redefined Assessment of Strength, Sensation and Prehension scores (GRASSP) | 48 months
  Change in baseline GRASSP results for strength, sensation and prehension at 48 months post-operatively. Five subtests: 1. Dorsal sensation (3 locations) each scored 0-4 (sum =subtest score, 0-12, with 0 being no sensation and 12 being normal sensation); 2. Palmar sensation (same as above); 3. Strength (10 muscles of arms and hand), motor grad 0-5 for each (sum = subtest total 0-50 with 0 being worst score and 50 being full motor function in all muscles); 4. Prehension ability - 3 grasps (cylindrical, lateral key, tip to tip) - each scored 0-4 (sum=subtest score, 0-12 with 0 being worst function and 12 being no dysfunction); 5 Prehension performance - 6 prehension tasks (pour water, open jars, pick up and turn key, transfer 9 pegs from board, pick up four coins and place in slot and screw 4 nuts on bolt - each scored 0-5 (sum=subtest score 0-30 with 0 being worst score to 30 being best possible score.
Neuro Quality of Life - Depression Short Form (NQOL-Dep) | 48 months
  Changes in baseline NQOL-Dep scores at 48 months post-operatively. Scores range from 8-40 with 8 being best outcome and 40 being the worst outcome
Neuro Quality of Life - Upper Extremity Short Form (NQOL-UEF) | 48 Months
  Changes in baseline NQOL-UEF scores at 48 months post-operatively. Scores range from 8-40 with 40 being the best outcome and 8 being the worst possible outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Z Ray, MD, Principal Investigator — Washington University School of Medicine
Locations (9):
- United States (7):
  - Stanford University, Stanford, California
  - University of Miami, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Houston Methodist, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - Alberta Health Services - Foothills Medical Center, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data. Only aggregate data will be published.

REFERENCES:
- See also: Washington University Neurosurgery Website — http://www.neurosurgery.wustl.edu